CLINICAL TRIAL: NCT06570317
Title: Prospective, Multicentre Phase II Clinical Study of Nintedanib for the Prevention of Radiation Pneumonia in Unresectable NSCLC
Brief Title: Nintedanib for the Prevention of Radiation Pneumonia in Unresectable NSCLC
Status: Recruiting | Type: Observational
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Gang Jin, Director, Second Hospital of Shanxi Medical University
Other Study IDs: [2024]YX No. 273
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: NSCLC; Nintedanib; Radiation Pneumonitis
MeSH Terms: conditions — Radiation Pneumonitis | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Nintedanib — For patients with unresectable NSCLC, nidanib is administered during sequential radiotherapy

SUMMARY:
This study is aimed at patients with unresectable NSCLC who take nintedanib during sequential radiotherapy to explore the incidence of radiation pneumonitis above grade 2 in the nintedanib combined with radiotherapy mode and observe safety. And will further explore the progression-free survival (PFS) and overall survival (OS) of patients treated with nintedanib in combination with radiotherapy and immunotherapy.

Primary objective: To evaluate the safety of nintedanib combined with sequential radiotherapy in patients with unresectable NSCLC and the incidence of radiation pneumonitis above grade 2. Secondary objective: To evaluate the changes in lung function, progression-free survival (PFS) and overall survival (OS) in patients with unresectable NSCLC after nintedanib combined with sequential radiotherapy.

Patients need to receive induction therapy, chemotherapy and/or immunotherapy for at least one cycle. Then they will receive sequential radiotherapy and nintedanib for 6 months. Finally, they will receive immunotherapy maintenance therapy for 16 cycles.

ELIGIBILITY:
Inclusion Criteria:

* 1) Men or women who are over 18 years old (including 18 years old) when signing the informed consent form;
* 2) Non-small cell lung cancer was confirmed by histology and could not be resected, and EGFR/ALK driver gene was confirmed negative by gene mutation examination;
* 3) At least one measurable lesion with imaging examination (according to RECIST1.1) is examined by spiral CT or MR, and the length and diameter of the lesion are ≥ 10 mm;
* 4) within 3 days before treatment, the score according to ECOG is 0 ~ 1;
* 5) Life expectancy ≥3 months;
* 6)The vital organs function well,
* 7)The subjects volunteered to join the study and signed the informed consent form, with good compliance and cooperation with the follow-up.

Exclusion Criteria:

* 1) Complicated with severe respiratory diseases: pulmonary fibrosis, active tuberculosis, etc.
* 2)Persons with mental disorder, blood system diseases, autoimmune diseases and serious primary diseases of heart, brain, liver and kidney;
* 3) Hemorrhagic events that require blood transfusion, invasive intervention or hospitalization occur within 3 months before the first administration, or there are bleeding symptoms and need intervention treatment (such as hemoptysis, hematuria and bloody stool), or high-risk factors with bleeding risk (such as tumor surrounding or invading important blood vessels, obvious necrosis or cavity around tumor, esophageal varices, etc.);
* 4) Thrombosis or embolic diseases, abnormal blood coagulation function and bleeding tendency;
* 5) Known or suspected to be allergic to the study drug and its auxiliary materials;
* 6) The baseline pregnancy test of pregnant and lactating women or fertile women is positive.
* 7) According to the researcher's judgment, the subjects have other factors that may lead to the forced termination of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men or women over the age of 18 (including 18 years old), whose vital organs function well, who are diagnosed as non-small cell lung cancer by histology and cannot be surgically removed, and whose EGFR/ALK driver gene is negative by gene mutation test. The score of physical fitness in the Eastern Cooperative Oncology Group (ECOG) is 0 ~ 1, and the life expectancy is ≥3 months. At least one measurable lesion (non-brain) according to RECISTv1.1.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-08-24 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
security | Up to 2 years
  Incidence of adverse events
Incidence rate of radiation pneumonia | Up to 2 years
  Incidence of grade 2 and above radiation pneumonia

SECONDARY OUTCOMES:
Pulmonary function index | Up to 2 years
  Changes of pulmonary function indexes（FEV1, Dlco）
Progression-free Survival (PFS) | Up to 2 years
  From the date of enrollment to the date of disease progression
Overall Survival (OS) | Up to 2 years
  From the date of enrollment until death by any cause or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, Dr., Principal Investigator — Second Hospital of Shanxi Medical University
Locations (7):
- China (7):
  - Jincheng General Hospital, Jincheng, Shanxi
  - Jinzhong third people's hospital, Jinzhong, Shanxi
  - Frist Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Hospital of Traditional Chinese Medicine, Taiyuan, Shanxi
  - TISCO General Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No